CLINICAL TRIAL: NCT02319941
Title: Comparison of Low-Dose, Standard-Dose Ticagrelor and Clopidogrel for Inhibition of Platelet Reactivity in Patients With Acute Coronary Syndromes; Pharmacodynamics and Pharmacokinetics Study
Brief Title: Comparison of Low-Dose, Standard-Dose Ticagrelor and Clopidogrel for Inhibition of Platelet Reactivity in Patients With Acute Coronary Syndromes
Acronym: OPTIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: AstraZeneca (Industry); Roche Pharma AG (Industry); KBM pharm (Unknown)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2014-07
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Inhibition of Platelet Reactivity; ticagrelor; clopidogrel; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose ticagrelor (Experimental): 60mg bid
  Interventions: Drug: ticagrelor
- standard dose ticagrelor (Active Comparator): 90mg bid
  Interventions: Drug: ticagrelor
- standard dose clopidogrel (Active Comparator): 75mg qd
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: ticagrelor
  Arms: Low dose ticagrelor; standard dose ticagrelor
Drug: clopidogrel
  Arms: standard dose clopidogrel

SUMMARY:
The purpose of this study is to compare Low-Dose, Standard-Dose Ticagrelor and Clopidogrel for Inhibition of Platelet Reactivity in Patients with Acute Coronary Syndromes

ELIGIBILITY:
Inclusion Criteria:

* ST elevation or non ST elevation acute coronary syndrome patients of chest pain within 24 hours

Exclusion Criteria:

* Known hypersensitivity to clopidogrel and ticagrelor and aspirin
* Treatment with anticoagulants
* Exposure to a thrombolytic agent within 24 hours prior to randomization
* Use of glycoprotein IIb - IIIa inhibitors at randomization
* History of major hemorrhage (intracranial, gastrointestinal, etc.)
* clotting disorder and/or bleeding disorder
* Any history of Severe renal or hepatic dysfunction
* Hematologic disorder including a Hemoglobin less than 10 g/L or a platelet count less than 80,000 cells/mm3
* Cardiac shock, severe left ventricular dysfunction LVEF less than 30%
* Sick sinus syndrome or second degree of av block without permanent pacemaker
* No concurrent cytochrome p450 3a inhibitors and enhancers within 2 weeks
* Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg,drug and alcohol abuse, mental illness) or that could prevent, limit, or confound the protocol-specified assessments.
* Life expectancy of less than 6 months
* Pregnancy or lactating
* Participation in any drug study in the previous 3 months
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
P2Y12 reaction units(PRU) | 8 hours and 30days after first randomized dose
  P2Y12 Reaction Units (PRU) measured by VerifyNow P2Y12 assay

SECONDARY OUTCOMES:
Percentage inhibition of platelet aggregation | 0, 0.5, 1, 2, 4, 8,24 hours and 30 days after first randomized study treatment
Aggregation units(AU), Area Under the Curve(AUC) | 0, 0.5, 1, 2, 4, 8,24 hours and 30 days after first randomized study treatment
  by Multiplate analyzer
Percentage of low-responsive patients | 0, 0.5, 1, 2, 4, 8,24 hours and 30 days after first randomized study treatment
  Low-responsive patients is defined as PRU ≥ 235 from VerifyNow P2Y12 and/or percentage of platelet inhibition <15%
Description of the pharmacokinetic (PK) profile for Ticagrelor and its metabolite AR-C124910XX | 0, 0.5, 1, 2, 4, 8, 10,24 hours after first randomized study treatment
  in terms of maximum concentration (Cmax),time to maximum concentration (tmax) and area under the concentration curve from time zero to infinity (AUC), t1/2, CL/F
MACE(Major adverse cardiac event) | 30 days after first randomized study treatment
  Death, Myocardial Infarction, stent thrombosis, stroke,
Adverse event | 30 days after first randomized study treatment
  including bleeding by TIMI/PLATO criteria, dyspnea, bradycardia, syncope,
Drug tolerance | 30 days after first randomized study treatment
  Drug tolerance is evaluated as adverse event following discontinuation of drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Park DW, Lee PH, Jang S, Lim HS, Kang DY, Lee CH, Ahn JM, Yun SC, Park SW, Park SJ. Effect of Low-Dose Versus Standard-Dose Ticagrelor and Clopidogrel on Platelet Inhibition in Acute Coronary Syndromes. J Am Coll Cardiol. 2018 Apr 10;71(14):1594-1595. doi: 10.1016/j.jacc.2018.02.010. No abstract available. PMID 29622168